CLINICAL TRIAL: NCT05653362
Title: A Randomized Trial Evaluating Coconut Oil as an Alternative to Commercial Ultrasound Gel in Obstetrical Ultrasounds
Brief Title: Coconut Oil vs. Commercial Ultrasound Gel In Obstetric Ultrasounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Caroline Rouse, Assistant professor of Obstetrics and Gynecology, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 12932
Record Dates: First submitted 2022-11-10; First posted 2022-12-16 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy, High Risk
Keywords: ultrasonography; coconut oil; ultrasound gel

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Coconut Oil followed by Commercial Ultrasound Gel (Other): After the patient is consented and all questions are answered, the patient's information will be entered into a RedCap and they will be randomized to either starting the scan by first obtaining the required study images with coconut oil and then proceeding to the standard ultrasound using commercial ultrasound gel (Arm 1) or to starting with the scheduled ultrasound using the commercial ultrasound gel and ending by obtaining the required study images using coconut oil (Arm 2).
  Whether assigned to Arm 1 or Arm 2, prior to the collection of the study images using coconut oil, the participant will be handed a small plastic cup with a pre-measured amount of coconut oil and they will be asked to warm it in their hand for at least 2 minutes. They will then apply the coconut oil to their own abdomen with their hands prior to the ultrasound technician obtaining the required images.
  The ultrasound technician will collect 3 extra images for study purposes only using the coconut oil.
  Interventions: Device: Coconut Oil; Device: Commercial Ultrasound Gel
- Commercial Ultrasound Gel followed by Coconut Oil (Other): After the patient is consented and all questions are answered, the patient's information will be entered into a RedCap and they will be randomized to either starting the scan by first obtaining the required study images with coconut oil and then proceeding to the standard ultrasound using commercial ultrasound gel (Arm 1) or to starting with the scheduled ultrasound using the commercial ultrasound gel and ending by obtaining the required study images using coconut oil (Arm 2).
  Whether assigned to Arm 1 or Arm 2, prior to the collection of the study images using coconut oil, the participant will be handed a small plastic cup with a pre-measured amount of coconut oil and they will be asked to warm it in their hand for at least 2 minutes. They will then apply the coconut oil to their own abdomen with their hands prior to the ultrasound technician obtaining the required images.
  The ultrasound technician will collect 3 extra images for study purposes only using the coconut oil.
  Interventions: Device: Coconut Oil; Device: Commercial Ultrasound Gel

INTERVENTIONS:
Device: Coconut Oil — Coconut oil was applied to the patients' abdomen during the ultrasound to serve as a conducting medium. When applied topically, coconut oil is not absorbed systemically by the subject and will not affect the fetus. There are no studies showing a potential risk of the use of topical coconut oil in pregnancy. Subjects with a coconut allergy will be excluded from this study due to risk of allergic reaction.
Device: Commercial Ultrasound Gel — Room-temperature Aquasonic 100 (Parker Laboratories, Inc., Fairfield, NJ) applied to patients' abdomen during the ultrasound to serve an another conducting medium.

SUMMARY:
The goal of this randomized controlled trial is to compare the use of coconut oil with commercial ultrasound gel for obstetrical ultrasounds. The main questions it aims to answer are:

1. To evaluate the quality of ultrasound images obtained using coconut oil compared with commercial ultrasound gel.
2. To access patient acceptability of coconut oil as compared to commercial ultrasound gel.

Participants will:

1. Allow a total of 6 study images to be obtained; 3 using coconut oil and 3 with commercial ultrasound gel.
2. Fill out a 10-question, 5-point Likert scale survey following their ultrasound with both coupling mediums to compare acceptability.

DETAILED DESCRIPTION:
After receiving institutional review board approval, we conducted a randomized 2x2 crossover study. Patients could be enrolled in the study if they had a singleton pregnancy and were presenting for a routine growth or anatomy ultrasound. Exclusion criteria included an allergy to coconut, active inflammatory dermatologic conditions, and a multiple gestation pregnancy. A single ultrasound machine (GE Voluson E10) was used to obtain all images during this study. The three standard fetal biometry views - biparietal diameter (BPD)/head circumference (HC), abdominal circumference (AC), and femur length (FL) - were obtained by qualified ultrasound technicians for each patient with both coupling agents, for a total of six study images per patient. After obtaining written consent, study data were collected and managed using REDCap electronic data capture tools. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources.

Patients were randomized to either starting their scheduled ultrasound exam by obtaining the three study images using coconut oil and then proceeding with the standard ultrasound using commercial ultrasound gel or vice versa. A total of 15g of room-temperature, organic, refined coconut oil was used for each patient. The commercial ultrasound gel used for this study was room-temperature Aquasonic 100 (Parker Laboratories, Inc., Fairfield, NJ) of an unmeasured amount. The patient's abdomen was cleaned off with a towel between applications of each coupling agent. After completion of the ultrasound session, patient satisfaction with both coupling agents was assessed using a ten-question acceptability survey measured on a five-point Likert scale which was adapted from a previously validated survey.

Using a quantifiable scale developed for this study (0-25: unacceptable, 26-50: suboptimal, 51-75: acceptable, and 76-100: optimal), two experienced Maternal-Fetal Medicine physicians rated all study images on quality, resolution, and detail as defined by prior studies2. Quality was defined as an overall assessment of the image encompassing contrast of solid and fluid-filled structures. Resolution was defined as the sharpness and crispness of the image as well as a lack of haziness/blurriness. Detail was defined as the clarity of landmarks and ease with which boundaries of structures are seen and how well they are defined. Using Viewpoint (GE Healthcare), an ultrasound viewing software, the six study images for each patient were presented in the order of coupling agent each patient was randomized to first and second. Each set of three images per coupling agent was in the following order: BPD/HC, AC, and FL. The physicians rating the images were blinded to the agent used to capture each image and had no knowledge of the randomization list created by the study statisticians.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Patients presenting for an anatomy or growth US
* Patients assigned to the pre-determined ultrasound suite that will stay constant throughout the study so that the same ultrasound machine is used to obtain all images.

Exclusion Criteria:

* Allergy to coconut
* Active inflammatory dermatologic conditions (dermatitis, eczema, or psoriasis)
* Multiple gestation pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Rouse, MD, Principal Investigator — Indiana University Department of Maternal Fetal Medicine
Locations (1):
- Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agero AL, Verallo-Rowell VM. A randomized double-blind controlled trial comparing extra virgin coconut oil with mineral oil as a moisturizer for mild to moderate xerosis. Dermatitis. 2004 Sep;15(3):109-16. doi: 10.2310/6620.2004.04006. PMID 15724344
- [Background] DebMandal M, Mandal S. Coconut (Cocos nucifera L.: Arecaceae): in health promotion and disease prevention. Asian Pac J Trop Med. 2011 Mar;4(3):241-7. doi: 10.1016/S1995-7645(11)60078-3. Epub 2011 Apr 12. PMID 21771462
- [Background] Kabara JJ, Swieczkowski DM, Conley AJ, Truant JP. Fatty acids and derivatives as antimicrobial agents. Antimicrob Agents Chemother. 1972 Jul;2(1):23-8. doi: 10.1128/AAC.2.1.23. PMID 4670656
- [Background] Esquenazi D, Wigg MD, Miranda MM, Rodrigues HM, Tostes JB, Rozental S, da Silva AJ, Alviano CS. Antimicrobial and antiviral activities of polyphenolics from Cocos nucifera Linn. (Palmae) husk fiber extract. Res Microbiol. 2002 Dec;153(10):647-52. doi: 10.1016/s0923-2508(02)01377-3. PMID 12558183

RESULTS

PARTICIPANT FLOW:
Groups:
- Coconut Oil Followed by Commercial Ultrasound Gel: This group obtained standard biometry ultrasound images first with coconut oil and then with commercial ultrasound gel.
- Commercial Ultrasound Gel Followed by Coconut Oil: This group obtained standard biometry ultrasound images first with commercial ultrasound gel and then with coconut oil.
Period: Overall Study
Arm/Group | Coconut Oil Followed by Commercial Ultrasound Gel | Commercial Ultrasound Gel Followed by Coconut Oil
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Coconut Oil Followed by Commercial Ultrasound Gel; Commercial Ultrasound Gel Followed by Coconut Oil: Patients could be enrolled if they had a singleton pregnancy and were presenting for a routine growth or anatomy ultrasound. Exclusion criteria included an allergy to coconut, active inflammatory dermatologic conditions, and a multiple gestation pregnancy. After obtaining written consent from study participants, data were collected and managed using REDCap electronic data capture tools. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies. A single ultrasound machine (GE Voluson E10) was used to obtain all images during this study. The three standard fetal biometry views - biparietal diameter (BPD)/head circumference (HC), abdominal circumference (AC), and femur length (FL) - were obtained by qualified ultrasound technicians for each patient with both coupling agents, for a total of six study images per patient.
  Patients were randomized to the sequence in which they would receive the coupling agents (i.e., either starting their scheduled ultrasound exam by obtaining the three study images using coconut oil and then proceeding with the standard ultrasound using commercial ultrasound gel or vice versa). Ultimately, forty patients were randomized into two even groups. Neither patients nor ultrasound technicians were blinded from sequence assignment, but physicians rating the images were blinded to assignment.
- Total: Total of all reporting groups
Arm/Group | Coconut Oil Followed by Commercial Ultrasound Gel | Commercial Ultrasound Gel Followed by Coconut Oil | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Data were not collected.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Quality of Ultrasound Images
Description: The quality of ultrasound images obtained using coconut oil compared with commercial ultrasound gel was assessed using a quantifiable scale developed for this study (0-25: unacceptable, 26-50: suboptimal, 51-75: acceptable, and 76-100: optimal). Using Viewpoint (GE Healthcare), an ultrasound viewing software, the six study images for each patient were presented in the order of coupling agent each patient was randomized to first and second. Each set of three images per coupling agent was in the following order: Biparietal Diameter/Head circumference (BPD/HC), abdominal circumference (AC), and femur length (FL). The physicians rating the images were blinded to the agent used to capture each image and had no knowledge of the randomization list created by the study statisticians. The image quality scores given by the two experienced Maternal-Fetal Medicine physicians were averaged to compute a single score for each image per coupling agent.
Time Frame: ultrasound scanning, an average of 1 hour
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Coconut Oil Quality; Commercial Ultrasound Gel Quality: Quality was defined as an overall assessment of the image encompassing contrast of solid and fluid-filled structures.
Arm/Group | Coconut Oil Quality | Commercial Ultrasound Gel Quality
Number analyzed (Participants) | 40 | 40
score on a scale
  BPD/HC | 76.05 (3.75) | 76.14 (3.75)
  AC | 75.18 (2.50) | 76.35 (2.50)
  FL | 78.00 (0.88) | 79.13 (0.88)

2. Secondary Outcome: Acceptability
Description: Patient acceptability of coconut oil as compared to commercial ultrasound gel was assessed using a ten-question acceptability survey measured on a five-point Likert scale which was adapted from a previously validated survey. Higher scores meant a better outcome for questions 1 and 2 and a lower score meant a better outcome for questions 3, 4, and 5. The minimum value was a score of 1 and the maximum value was a score of 5.
Time Frame: after ultrasound scanning, an average of 1 hour
Population: The arms/groups are combined because each participant had images obtained with both coconut oil and standard ultrasound gel during their ultrasound. It was only the order of application that was randomized so as not to bias the acceptability survey. Data was collected after every participant had all images obtained (4 with coconut oil and 4 with standard gel), not separately after each application.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Coconut Oil Followed by Commercial Ultrasound Gel: Patients had obstetric ultrasound done with coconut oil prior to commercial ultrasound gel.
- Commercial Ultrasound Gel Followed by Coconut Oil: Patients had obstetric ultrasound done with commercial ultrasound gel prior to coconut oil.
Arm/Group | Coconut Oil Followed by Commercial Ultrasound Gel | Commercial Ultrasound Gel Followed by Coconut Oil
Number analyzed (Participants) | 20 | 20
units on a scale
  The gel/coconut oil used in the scan was messy. | 4.08 (4) | 2.55 (2)
  I experienced itching/burning/redness from the scan. | 4.83 (5) | 4.65 (5)
  The gel/coconut oil was easy to remove/rub in after the scan. | 4.50 (5) | 3.48 (4)
  I like how my skin felt after using the gel/coconut oil. | 4.55 (4) | 2.70 (3)
  I would have a scan with this gel again. | 4.68 (4) | 3.78 (4)

ADVERSE EVENTS:
Time Frame: ultrasound scanning, an average of 1 hour
Groups:
- Coconut Oil: All participants were exposed to coconut oil at some point during the study.
- Ultrasound Gel: All participants were exposed to ultrasound gel at some point during the study.
Arm/Group | Coconut Oil | Ultrasound Gel
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
Technicians and patients were not blinded. This study was performed at a single site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT05653362/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT05653362/ICF_001.pdf